CLINICAL TRIAL: NCT05598203
Title: Effect of Nutritional Education Groups Added in the Usual Care of Outpatients with Type 2 Diabetes: a Randomized Clinical Trial
Brief Title: Effect of Nutrition Education Groups in the Treatment of Patients with Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20220238
Record Dates: First submitted 2022-10-13; First posted 2022-10-28 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Glycated Hemoglobin A; Food and Nutrition Education; Feeding Behavior; Diabetes Complications; Body Mass Index; Lipids; Blood Pressure; Outcome Assessment, Health Care
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Feeding Behavior; Diabetes Complications

STUDY DESIGN:
Intervention Model Description: Each group will be exposed to only one of the factors, diabetes education operative groups added usual individual counseling; or usual individual counseling.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive four group meetings in addition to the usual care, specifically in the form of operative groups. Participants in these groups will actively participate in the sessions and will be given tasks to complete at home. There will be four sessions, which can be held weekly, fortnightly or monthly, depending on the availability of participants. Each participant will attend each meeting only once. These sessions, lasting one hour, will take place at the Hospital de Clínicas de Porto Alegre and approximately 20 participants will be invited to each group.
  Topics covered in these sessions will include:
  1. "Let's go shopping" = purchasing food through NOVA classification and nutritional labeling and food labels
  2. "Healthy Plate" = Diabetes Plate Method.
  3. "Hunger and satiety" = signs of hunger and satiety and eating mindfully
  Interventions: Behavioral: Operative group of nutrition education
- Control (usual treatment) (Active Comparator): In the usual care provided, there will be a consultation with a dietitian every four months. This consultation will involve nutritional counseling, where up to five combinations of lifestyle changes will be agreed upon with the participant. The combinations will be tailored to individual needs and align with diabetes recommendations, emphasizing increased consumption of natural foods, organizing meals according to the Diabetes Plate method, and promoting a reduction in sedentary time. Subsequent visits will reassess the combinations of lifestyle changes, addressing barriers and motivations identified during the counseling process.
  Patients will not be encouraged to implement caloric restrictions, but they will be motivated to adopt healthy eating patterns in accordance with the recommendations of the American Diabetes Association and the Sociedade Brasileira de Diabetes.
  Interventions: Behavioral: Operative group of nutrition education

INTERVENTIONS:
Behavioral: Operative group of nutrition education — The intervention will be carried out with operational nutritional education groups. Four meetings will be held, each meeting lasting one hour, weekly or fortnightly (according to the availability of the patient). The following foods proposed foods: Meeting 1 = education on classification labels and proposed foods proposed foods (education on classification labels and substitution of Brazilian foods), in this guide meeting the proposal is processed or ultra-processed by an in natura food or minimally processed; Meeting 2 = assembly of the healthy dish (food portions, food index and glycemic load, food clothes), the proposal in this meeting is the assembly of the complete dish in the meals eaten throughout the day; and Encounter 3 = hunger and satiety (aiming to increase the perception of hunger and satiety signals), encounter as a task to be accomplished; Encounter 4 = strengthening change, barriers and difficulties in maintaining habits based on the transtheoretical model of change.

SUMMARY:
Every year there is an increase in people with diabetes all over the world. Because it is a disease associated with several comorbidities and is increasing, there is a need for more effective treatments. Lifestyle changes combined with medication are the best strategies for the treatment and reduction of comorbidities. Therefore, the present study posits the hypothesis that the integration of nutritional education groups into standard treatment, within a nutrition-specialized outpatient clinic, may yield additional enhancements in health parameters among patients diagnosed with type 2 diabetes. The driving force behind this research lies in the pursuit of more effective strategies to enhance glycemic control, diminish the risk of complications, and elevate the overall quality of life for these patients. Our motivation stems from a commitment to base our interventions on scientific evidence and strive towards meaningful improvements in diabetes management outcomes. A randomized clinical trial will be conducted with adult patients with a previous diagnosis of type 2 diabetes. Patients will be divided into two groups (intervention: nutritional education added the usual care; and control: usual care). The outcomes analyzed will be: glycemic control, lipid profile, body mass and dynapenia obesity, blood pressure values, eating behavior, diabetes complications and adherence to recommendations.

DETAILED DESCRIPTION:
The estimate of patients with diabetes increases every year and for their treatment, a change in lifestyle is essential, so there is a need to seek strategies that increase patient adherence in the long term. Therefore, the present study posits the hypothesis that the integration of nutritional education groups into standard treatment, within a nutrition-specialized outpatient clinic, may yield additional enhancements in health parameters among patients diagnosed with type 2 diabetes. The driving force behind this research lies in the pursuit of more effective strategies to enhance glycemic control, diminish the risk of complications, and elevate the overall quality of life for these patients. Our motivation stems from a commitment to base our interventions on scientific evidence and strive towards meaningful improvements in diabetes management outcomes.

An open randomized clinical trial will be performed. Patients = patients with type 2 DM; Intervention = food (nutritional) education based on operative groups added the usual care; Control = usual care; Outcome/Outcomes = glycemic control, lipid profile, body mass and dynapenia obesity, blood pressure values, eating behavior, diabetes complications and adherence to recommendations. In order to detect a mean difference of 0.59 in HbA1c between patients randomized to the intervention (patient-centered group) and those in the control group (traditional education intervention), with a standard deviation of 1.39%, a type I error of 5%, and a type II error of 20%, a total of 88 patients in each group were deemed necessary (1:1 ratio at randomization, n= 176). Considering a dropout rate of 30% over the long term (12 months), it will be essential to include a total of 252 participants.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients with a previous diagnosis of type 2 diabetes mellitus

Exclusion Criteria:

* Patients with other types of diabetes
* With HbA1C within the therapeutic target or with values greater than 12%
* Severe neuropathy
* Chronic kidney disease [glomerular filtration rate <30mL/min/1.73m²]
* Life expectancy <6 months
* Chemical dependence/alcoholism or use of antipsychotics
* Autoimmune disease or chronic steroid use
* Gastroparesis
* Pregnant or lactating women
* Patients who have had an Episode of Acute Coronary Syndrome (ACS) in the last 60 days
* Wheelchair users
* Cognitive, neurological or psychiatric condition

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in baseline HbA1C at 4 months | From baseline to 4 months
  The Glycated Hemoglobin test (high precision chromatography on a Merck-Hitachi 9100 device with reference values of 4.8-6.0%) will be performed at the Clinical Pathology Laboratory of the Hospital de Clínicas de Porto Alegre (HCPA) by means of blood sample. The patient will be instructed to fast for 12 hours.
Change in baseline HbA1C at 8 months | From baseline to 8 months
  The Glycated Hemoglobin test (high precision chromatography on a Merck-Hitachi 9100 device with reference values of 4.8-6.0%) will be performed at the Clinical Pathology Laboratory of the Hospital de Clínicas de Porto Alegre (HCPA) by means of blood sample. The patient will be instructed to fast for 12 hours.
Change in baseline HbA1C at 12 months | From baseline to 12 months
  The Glycated Hemoglobin test (high precision chromatography on a Merck-Hitachi 9100 device with reference values of 4.8-6.0%) will be performed at the Clinical Pathology Laboratory of the Hospital de Clínicas de Porto Alegre (HCPA) by means of blood sample. The patient will be instructed to fast for 12 hours.
Change in diabetic retinopathy and baseline diabetic kidney disease at 12 months | From baseline to 12 months
  Diabetes kidney disease and diabetic retinopathy will be collected from patients' electronic medical records at baseline and at the end of the study (12 months).

SECONDARY OUTCOMES:
Change in basal body mass index at 4 months | From baseline to 4 months
  Anthropometric measurements will be used to assess nutritional status and will include weight (with light clothes and without shoes) and height. For such measurements, an anthropometric scale and a fixed wall stadiometer will be used. BMI will be calculated from the formula weight (kg)/height2) and will be considered healthy weight (therapeutic target) when <25 kg/m2 for adults and <27 kg/m2 for the elderly.
Change in basal body mass index at 8 months | From baseline to 8 months
  Anthropometric measurements will be used to assess nutritional status and will include weight (with light clothes and without shoes) and height. For such measurements, an anthropometric scale and a fixed wall stadiometer will be used. BMI will be calculated from the formula weight (kg)/height2) and will be considered healthy weight (therapeutic target) when <25 kg/m2 for adults and <27 kg/m2 for the elderly.
Change in basal body mass index at 12 months | From baseline to 12 months
  Anthropometric measurements will be used to assess nutritional status and will include weight (with light clothes and without shoes) and height. For such measurements, an anthropometric scale and a fixed wall stadiometer will be used. BMI will be calculated from the formula weight (kg)/height2) and will be considered healthy weight (therapeutic target) when <25 kg/m2 for adults and <27 kg/m2 for the elderly.
Change in basal metabolic control at 4 months | From baseline to 4 months
  The analyzes will be carried out at the Clinical Pathology Laboratory of the Hospital de Clínicas de Porto Alegre and will comprise: fasting plasma glucose (measured by the enzymatic glucose-peroxidase method - Biodiagnostic Kit), total cholesterol (colorimetric enzymatic method), HDL cholesterol (colorimetric reaction enzyme analysis, methods described by Farish and modified Fletcher) and serum triglycerides (colorimetric enzymatic method using a commercial kit, as described by McGowan). LDL cholesterol will be calculated using the Friedewald formula for patients with serum triglycerides below 400 mg/dL. The patient will be instructed to fast for 12 hours. Fasting glucose values between 80 - 130 mg/dL, HbA1c <7%, LDL-cholesterol <100 mg/dL and triglycerides <150 mg/dL will be considered within the recommended therapeutic target. Patients with HbA1c <7.0% (adults) and <7.5% (elderly) will be considered with good glycemic control.
Change in basal metabolic control at 8 months | From baseline to 8 months
  The analyzes will be carried out at the Clinical Pathology Laboratory of the Hospital de Clínicas de Porto Alegre and will comprise: fasting plasma glucose (measured by the enzymatic glucose-peroxidase method - Biodiagnostic Kit), total cholesterol (colorimetric enzymatic method), HDL cholesterol (colorimetric reaction enzyme analysis, methods described by Farish and modified Fletcher) and serum triglycerides (colorimetric enzymatic method using a commercial kit, as described by McGowan). LDL cholesterol will be calculated using the Friedewald formula for patients with serum triglycerides below 400 mg/dL. The patient will be instructed to fast for 12 hours. Fasting glucose values between 80 - 130 mg/dL, HbA1c <7%, LDL-cholesterol <100 mg/dL and triglycerides <150 mg/dL will be considered within the recommended therapeutic target. Patients with HbA1c <7.0% (adults) and <7.5% (elderly) will be considered with good glycemic control.
Change in basal metabolic control at 12 months | From baseline to 12 months
  The analyzes will be carried out at the Clinical Pathology Laboratory of the Hospital de Clínicas de Porto Alegre and will comprise: fasting plasma glucose (measured by the enzymatic glucose-peroxidase method - Biodiagnostic Kit), total cholesterol (colorimetric enzymatic method), HDL cholesterol (colorimetric reaction enzyme analysis, methods described by Farish and modified Fletcher) and serum triglycerides (colorimetric enzymatic method using a commercial kit, as described by McGowan). LDL cholesterol will be calculated using the Friedewald formula for patients with serum triglycerides below 400 mg/dL. The patient will be instructed to fast for 12 hours. Fasting glucose values between 80 - 130 mg/dL, HbA1c <7%, LDL-cholesterol <100 mg/dL and triglycerides <150 mg/dL will be considered within the recommended therapeutic target. Patients with HbA1c <7.0% (adults) and <7.5% (elderly) will be considered with good glycemic control.
Change in baseline blood pressure at 4 months | From baseline to 4 months
  Three blood pressure measurements will be performed with a Digital Blood Pressure Monitor Omron sphygmomanometer model HEM-705CP, with an interval of one minute, with the patient sitting down after five minutes of rest, using a cuff of the appropriate size for the arm diameter.
Change in baseline blood pressure at 8 months | From baseline to 8 months
  Three blood pressure measurements will be performed with a Digital Blood Pressure Monitor Omron sphygmomanometer model HEM-705CP, with an interval of one minute, with the patient sitting down after five minutes of rest, using a cuff of the appropriate size for the arm diameter.
Change in baseline blood pressure at 12 months | From baseline to 12 months
  Three blood pressure measurements will be performed with a Digital Blood Pressure Monitor Omron sphygmomanometer model HEM-705CP, with an interval of one minute, with the patient sitting down after five minutes of rest, using a cuff of the appropriate size for the arm diameter.

OTHER OUTCOMES:
Change in baseline eating behavior at 4 months | From baseline to 4 months
  Eating behavior will be evaluated using the Intuitive Eating Scale-2 (IES-2), adapted to Portuguese. This scale, based on principles of intuitive eating, encompasses questions about food attitudes and has been designed to assess adherence to hunger and satiety signals. Food consumption will be estimated through the 24-hour dietary recalls Multiple-Pass Method. Additionally, the study will assess the frequency of consumption of sweets, sugary drinks, alcoholic beverages, fried foods, cooking oil, and added oil after preparation (specifying type and quantity per capita), as well as sausages, canned goods, preserves, industrialized seasonings, meat, and eggs.
Change in baselineeating behavior at 8 months | From baseline to 8 months
  Eating behavior will be evaluated using the Intuitive Eating Scale-2 (IES-2), adapted to Portuguese. This scale, based on principles of intuitive eating, encompasses questions about food attitudes and has been designed to assess adherence to hunger and satiety signals. Food consumption will be estimated through the 24-hour dietary recalls Multiple-Pass Method. Additionally, the study will assess the frequency of consumption of sweets, sugary drinks, alcoholic beverages, fried foods, cooking oil, and added oil after preparation (specifying type and quantity per capita), as well as sausages, canned goods, preserves, industrialized seasonings, meat, and eggs.
Change in baseline eating behavior at 12 months | From baseline to 12 months
  Eating behavior will be evaluated using the Intuitive Eating Scale-2 (IES-2), adapted to Portuguese. This scale, based on principles of intuitive eating, encompasses questions about food attitudes and has been designed to assess adherence to hunger and satiety signals. Food consumption will be estimated through the 24-hour dietary recalls Multiple-Pass Method. Additionally, the study will assess the frequency of consumption of sweets, sugary drinks, alcoholic beverages, fried foods, cooking oil, and added oil after preparation (specifying type and quantity per capita), as well as sausages, canned goods, preserves, industrialized seasonings, meat, and eggs.
Change in baseline dynapenia obesity at 4 months | From baseline to 4 months
  The SARC-F questionnaire (a simple tool for rapid sarcopenia diagnosis) will be administered by phone. Calf circumference will be measured at the point of greatest horizontal circumference, with the subject sitting, legs in a non-contracted position, and 20 cm apart. Handgrip strength will be assessed using a Hydraulic Hand Dynamometer (in the dominant hand), and the walking test will involve the patient walking a pre-marked distance of four meters (measured with the aid of a stopwatch). The cutoff points employed to identify low muscle strength will be <26 kg for men and <16 kg for women, with altered waist circumference defined as >102 for men and >88 for women. For dynapenic abdominal obesity, individuals with both low muscle strength and altered waist circumference will be considered.
Change in baseline dynapenia obesity at 8 months | From baseline to 8 months
  The SARC-F questionnaire (a simple tool for rapid sarcopenia diagnosis) will be administered by phone. Calf circumference will be measured at the point of greatest horizontal circumference, with the subject sitting, legs in a non-contracted position, and 20 cm apart. Handgrip strength will be assessed using a Hydraulic Hand Dynamometer (in the dominant hand), and the walking test will involve the patient walking a pre-marked distance of four meters (measured with the aid of a stopwatch). The cutoff points employed to identify low muscle strength will be <26 kg for men and <16 kg for women, with altered waist circumference defined as >102 for men and >88 for women. For dynapenic abdominal obesity, individuals with both low muscle strength and altered waist circumference will be considered.
Change in baseline dynapenia obesity at 12 months | From baseline to 12 months
  The SARC-F questionnaire (a simple tool for rapid sarcopenia diagnosis) will be administered by phone. Calf circumference will be measured at the point of greatest horizontal circumference, with the subject sitting, legs in a non-contracted position, and 20 cm apart. Handgrip strength will be assessed using a Hydraulic Hand Dynamometer (in the dominant hand), and the walking test will involve the patient walking a pre-marked distance of four meters (measured with the aid of a stopwatch). The cutoff points employed to identify low muscle strength will be <26 kg for men and <16 kg for women, with altered waist circumference defined as >102 for men and >88 for women. For dynapenic abdominal obesity, individuals with both low muscle strength and altered waist circumference will be considered.
Change in baseline adherence to recommendations at 4 months | From baseline to 4 months
  We will assess adherence to the nutritional combinations during each scheduled visit (at four, eight, and 12 months), as well as adherence to the Diabetes Plate Method. Additionally, the attendance of participants randomized to the intervention group will be monitored through their presence at the scheduled meetings, considering patients who attend at least two meetings. In the control group, assiduity will be evaluated based on return consultation attendance.
Change in baseline adherence to recommendations at 8 months | From baseline to 8 months
  We will assess adherence to the nutritional combinations during each scheduled visit (at four, eight, and 12 months), as well as adherence to the Diabetes Plate Method. Additionally, the attendance of participants randomized to the intervention group will be monitored through their presence at the scheduled meetings, considering patients who attend at least two meetings. In the control group, assiduity will be evaluated based on return consultation attendance.
Change in baseline adherence to recommendations at 12 months | From baseline to 12 months
  We will assess adherence to the nutritional combinations during each scheduled visit (at four, eight, and 12 months), as well as adherence to the Diabetes Plate Method. Additionally, the attendance of participants randomized to the intervention group will be monitored through their presence at the scheduled meetings, considering patients who attend at least two meetings. In the control group, assiduity will be evaluated based on return consultation attendance.

CONTACTS AND LOCATIONS:
Overall Officials: Jussara C De Almeida, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (2):
- Brazil (2):
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Universidade Federal do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul

REFERENCES:
- [Derived] Busanello A, Menezes VM, Koller OG, Volz Andreia A, de Almeida JC. Effect of group-based nutritional education combined with individual standard care for outpatients with type 2 diabetes: study protocol for a randomized clinical trial 1. Trials. 2025 Mar 6;26(1):78. doi: 10.1186/s13063-025-08720-1. PMID 40050966